CLINICAL TRIAL: NCT01824173
Title: Regulation of Muscle ATP Synthase Beta Subunit Metabolism in Obesity
Brief Title: Muscle Protein Metabolism in Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori R. Roust, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-004000
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: muscle; mitochondria; amino acids; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Amino Acid Infusion in Lean (Experimental): Amino Acid Infusion in Lean
  Interventions: Other: Increase in the levels of plasma amino acids
- Amino acid Infusion in Obese (Experimental): Amino acid Infusion in Obese
  Interventions: Other: Increase in the levels of plasma amino acids
- Exercise in lean (Experimental): Exercise in lean
  Interventions: Other: Aerobic exercise
- Exercise in Obese (Experimental): Exercise in Obese
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Increase in the levels of plasma amino acids — Aminosyn 15%; 160 mg/kg FFM/h for 4 hours
  Arms: Amino Acid Infusion in Lean; Amino acid Infusion in Obese
Other: Aerobic exercise — Moderate intensity for 45 minutes
  Arms: Exercise in Obese; Exercise in lean

SUMMARY:
Obesity is associated with reduced adenosine triphosphate (ATP) turnover in skeletal muscle, a condition that can impair muscle metabolism. The proposed research will discover mechanisms responsible for decreased content in mitochondrial proteins as well as in protein β-F1-ATPase, which is directly responsible for ATP assembly, in the muscle of obese individuals. This research will further examine the effectiveness of interventions, such as increased plasma amino acid availability and exercise, to increase the rate of production of mitochondrial proteins as well as that of β-F1-ATPase in the muscle of obese individuals. The findings will help to develop appropriate interventions to improve muscle ATP turnover and metabolism in obese people.

ELIGIBILITY:
Inclusion criteria:

1. Body mass index (BMI): lean, 19-26 kg/m2; obese, 30-40 kg/m2
2. Availability of transportation
3. Ability to sign informed consent form

Exclusion criteria:

1. Medication or supplements (i.e. amino acids, protein) known to affect protein metabolism
2. Presence of acute illness
3. History of liver disease
4. Uncontrolled metabolic disease
5. ECG documented abnormalities, atrial fibrillation, history of syncope, limiting or unstable angina, or congestive heart failure
6. Chronically elevated blood pressure (systolic, >140 mmHg; diastolic, >100 mmHg)
7. Cardiac pacemaker or other medical device implanted in the body
8. Low hemoglobin or hematocrit
9. Current participation in a weight-loss regimen, including extreme dietary practices
10. Smoking
11. Use of anabolic steroids or corticosteroids (within 3 months)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Rate of synthesis of muscle proteins (mixed muscle proteins, mitochondrial proteins, β-F1-ATPase) | Measured during a 9-hour infusion study

SECONDARY OUTCOMES:
β-F1-ATPase mRNA expression; PGC-1 expression | Measured during a 9-hour infusion study

CONTACTS AND LOCATIONS:
Overall Officials: Lori Roust, MD, Principal Investigator — Mayo Clinic; Christos S Katsanos, PhD, Principal Investigator — Arizona State University/Mayo Clinic Arizona
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Serrano N, Tran L, Hoffman N, Roust L, De Filippis EA, Carroll CC, Patel SH, Kras KA, Buras M, Katsanos CS. Lack of Increase in Muscle Mitochondrial Protein Synthesis During the Course of Aerobic Exercise and Its Recovery in the Fasting State Irrespective of Obesity. Front Physiol. 2021 Aug 2;12:702742. doi: 10.3389/fphys.2021.702742. eCollection 2021. PMID 34408662
- [Derived] Kras KA, Langlais PR, Hoffman N, Roust LR, Benjamin TR, De Filippis EA, Dinu V, Katsanos CS. Obesity modifies the stoichiometry of mitochondrial proteins in a way that is distinct to the subcellular localization of the mitochondria in skeletal muscle. Metabolism. 2018 Dec;89:18-26. doi: 10.1016/j.metabol.2018.09.006. Epub 2018 Sep 22. PMID 30253140
- [Derived] Tran L, Kras KA, Hoffman N, Ravichandran J, Dickinson JM, D'Lugos A, Carroll CC, Patel SH, Mandarino LJ, Roust L, Katsanos CS. Lower Fasted-State but Greater Increase in Muscle Protein Synthesis in Response to Elevated Plasma Amino Acids in Obesity. Obesity (Silver Spring). 2018 Jul;26(7):1179-1187. doi: 10.1002/oby.22213. Epub 2018 Jun 12. PMID 29896930
- [Derived] Kras KA, Hoffman N, Roust LR, Patel SH, Carroll CC, Katsanos CS. Plasma Amino Acids Stimulate Uncoupled Respiration of Muscle Subsarcolemmal Mitochondria in Lean but Not Obese Humans. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4515-4525. doi: 10.1210/jc.2017-01201. PMID 29029131
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials